CLINICAL TRIAL: NCT00684281
Title: Early Diagnosis of Alzheimer's Disease: Clinical, Neuropsychological and Neuroimaging Follow-up of a Cohort of Patients With an Isolated Memory Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-A00851-52; 2007-27
Record Dates: First submitted 2008-05-21; First posted 2008-05-26 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Magnetic Resonance Spectroscopy; DNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Subject control
  Interventions: Other: Neurological and neuropsychological consultation, MRI
- 2 (Experimental): 40 patients before hand include in a program
  Interventions: Other: Neurological and neuropsychological consultation, MRI, Studies in imaging of drip, DNA

INTERVENTIONS:
Other: Neurological and neuropsychological consultation, MRI — Neurological and neuropsychological consultation, MRI for the month 0, 18 and 36
  Arms: 1
Other: Neurological and neuropsychological consultation, MRI, Studies in imaging of drip, DNA — Neurological and neuropsychological consultation, MRI, Studies in imaging of drip, DNA, months 0/18/36
  Arms: 2

SUMMARY:
The aim of this project is to follow cohort of patients with aMCI in order to establish whether there are distinct subgroups in terms of evolution or aetiology, with distinct memory profiles and profiles of mesiotemporal atrophy and metabolic change

DETAILED DESCRIPTION:
The syndrome of "amnestic Mild Cognitive Impairment" (aMCI) has been introduced for patients with intact activities of daily living, with a memory complaint and objective memory decline on neuropathological assessment, without significative change in other domains of cognition. Follow-up in these patients shows that the memory impairment may remain stable or improve, while it worsens or extends to other cognitive domains in others, indicating prodromal AD.

ELIGIBILITY:
Inclusion Criteria:

* Patients beforehand include in the PHRC 2001 study (These patients presented to the inclusion in the PHRC 2001 a qualified board of amnestic Mild Cognitive Impairment [aMCI] or light cognitive confusion of type amnestic)
* The patient must be affiliated to an insurance scheme disease to participate in this study

Exclusion Criteria:

* For the magnetic resonance imaging: usual contraindications for an examination by MRI: claustrophobia, metal foreign bodies, pacemakers, etc.
* Incapacitated to realize the neuropsychological evaluation because of medical intercurrentes disorders
* Appointment of a guardian

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-07; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pursue the longitudinal study of a troop of subjects presenting an amnestic MCI in 36 months after the initial diagnosis | 36 months
Characterize the clinical evolution of these subjects: escalation with appearance of an insanity (of type Alzheimer's disease or of another type: degenerations fronto-temporal, insanity with body of Lewy), stabilization even improvement. | 36 months
Identify the neuropsychological markers and of neuroimaging structural and metabolic useful in clinical practice which allow to predict an escalation | 36 months
Identify the neuropsychological markers and of neuroimaging structural and metabolic useful in clinical practice which allow to predict a stabilization or an improvement. | 36 months
Improve the state of the knowledge on the origin of the confusions mnésiques isolated at the persons of fifty and more years old. | 36 months

SECONDARY OUTCOMES:
Establish diagnostic criteria which allow to improve the sensibility and the specificity of the premature diagnosis of MY. | 36 months
Determine if the ultra-premature diagnosis of MY at a stage where the hurts are still confined in the structures under - hippocampiques is possible. | 36 months
Determine the specific character or not of the infringement of the memory of visual recognition in the novice Alzheimer's disease. | 36 months
Determine the specific character or not the atrophy and the metabolic modifications of regions under - hippocampiques in the novice Alzheimer's disease. | 36 months
Inform the existence of process of functional compensation in the population of aMCI, notably to those who show themselves stable or improve. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu CECCALDI, MD, Principal Investigator — Assistance Publique des Hopitaux de Marseille
Locations (1):
- Hopital de la Timone- Service de neurologie et de neuropsychologie, Marseille, France